CLINICAL TRIAL: NCT03671733
Title: Effects of GLP-1 RAs on Weight and Metabolic Indicators in Obese Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201806897
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Liraglutide; Exenatide; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Liraglutide (Experimental): Administered subcutaneously (s.c., under the skin) once daily for 12 weeks.
  Interventions: Drug: Liraglutide
- Exenatide (Experimental): Administered subcutaneously (s.c., under the skin) twice daily for 12 weeks.
  Interventions: Drug: Exenatide
- Exenatide Microspheres for Injection (Experimental): Administered subcutaneously (s.c., under the skin) once weekly for 12 weeks.
  Interventions: Drug: Exenatide Microspheres for Injection

INTERVENTIONS:
Drug: Liraglutide — The treatment of Liraglutide lasted three months,During the first week: 0.6mg per day, subcutaneous injection;During the second week: 1.2mg per day, subcutaneous injection; From third week onwards, 1.8mg per day, subcutaneous injection.
  Other Names: Victoza
  Arms: Liraglutide
Drug: Exenatide — 10mcg once a day for 4 weeks increased to 10mcg twice a day for 8 weeks.
  Other Names: Byetta
  Arms: Exenatide
Drug: Exenatide Microspheres for Injection — Exenatide 2 mg injection once weekly for 12 weeks.
  Other Names: Bydureon
  Arms: Exenatide Microspheres for Injection

SUMMARY:
This studay evaluates the effect of the glucagon-like peptide-1 (GLP-1) receptor agonist,including Liraglutide,Exenatide and Exenatide Microspheres for Injection,in the treatment of subjects who are overweight or obese.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 65 years (to the date of screening)；
2. The newly diagnosed obese patients (BMI greater than 28 kg/m2) or abdominal obesity (male waist circumference is greater than 90cm, female waist is greater than 85cm).
3. Nearly a month have not used weight-related drugs,including various weight-loss drugs,GLP-1 analogs or agonists,metformin, acarbose,insulin,anti hyperthyroid drugs,etc;Or recently used weight-related drugs but the stable dose was more than 1 month,and the drug dose remained constant or decreased during the trial.
4. Weight stable for more than 3 months (weight fluctuations <5%).

Exclusion Criteria:

1. pregnant female.
2. Secondary diseases caused by other diseases: including hypothyroidism, increased cortisol, hypothalamic and pituitary lesions caused by obesity, all kinds of drug-induced obesity, and others.
3. Severe cardiovascular and cerebrovascular diseases (heart failure, myocardial infarction, acute hemorrhagic or ischemic encephalopathy), pulmonary heart disease or pulmonary insufficiency, renal failure, severe hepatitis.
4. Combined with acute complications of diabetes such as ketoacidosis, lactic acidosis, hyperosmolar state of diabetes.
5. Nearly a month had surgery, trauma, infection and so on.
6. Limb deformity incomplete, difficult to accurately determine the height, weight and other physical indicators.
7. Poor medication compliance or serious side effects (severe rash, syncope, etc.).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Weight Change at 3 months | baseline , 3 months
  Measured in kilograms

SECONDARY OUTCOMES:
Change in waist circumference | baseline and 3 months
  Measured in cm
Change in systolic blood pressure | baseline and 3 months
  Measured in mmHg
Change in diastolic blood pressure | baseline and 3 months
  Measured in mmHg
Change in HbA1c | baseline and 3 months
  Measured in %
Change in plasma glucose | baseline and 3 months
  Measured in mmol/l
Change in insulin | baseline and 3 months
  Measured in μU/ml
Change in lipids-total cholesterol | baseline and 3 months
  Measured in mmol/l
Change in lipids-low density lipoprotein cholesterol | baseline and 3 months
  Measured in mmol/l
Change in lipids-high density lipoprotein cholesterol | baseline and 3 months
  Measured in mmol/l
Change in lipids-triglycerides | baseline and 3 months
  Measured in mmol/l
Change in lipids-free fatty acids | baseline and 3 months
  Measured in μmol/l
Change in Uric Acid | baseline and 3 months
  Measured in mmol/l
Change in interleukin-6 | baseline and 3 months
  Measured in mmol/l
Change in tumor necrosis factor | baseline and 3 months
  Measured in mmol/l

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China